CLINICAL TRIAL: NCT04534205
Title: An Open-label Phase II/III Randomized Trial of BNT113 in Combination With Pembrolizumab Versus Pembrolizumab Monotherapy as a First Line Therapy in Patients With Unresectable Recurrent, or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) Which is Positive for Human Papilloma Virus 16 (HPV16+) and Expresses PD-L1
Brief Title: A Clinical Trial Investigating the Safety, Tolerability, and Therapeutic Effects of BNT113 in Combination With Pembrolizumab Versus Pembrolizumab Alone for Patients With a Form of Head and Neck Cancer Positive for Human Papilloma Virus 16 and Expressing the Protein PD-L1
Acronym: AHEAD-MERIT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT113-01; 2020-001400-41 (EudraCT Number); 2024-512671-12-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Unresectable Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Cancer; Recurrent Head and Neck Cancer
Keywords: Cancer vaccine; RNA vaccine; HNSCC; BNT113; Pembrolizumab; HPV16; Metastatic; Unresectable; Recurrent; Head and neck; mRNA vaccine; HPV-positive; Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Safety Run-In) - BNT113 + Pembrolizumab (Experimental): Safety Run-In Phase to confirm the safety and tolerability at the selected dose range level of BNT113 in combination with pembrolizumab.
  Interventions: Biological: BNT113; Biological: Pembrolizumab
- Part B (Randomized phase) - BNT113 + Pembrolizumab (Experimental): BNT113 in combination with pembrolizumab.
  Interventions: Biological: BNT113; Biological: Pembrolizumab
- Part B (Randomized phase) - Pembrolizumab monotherapy (Active Comparator): Pembrolizumab monotherapy.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: BNT113 — IV injection
  Arms: Part A (Safety Run-In) - BNT113 + Pembrolizumab; Part B (Randomized phase) - BNT113 + Pembrolizumab
Biological: Pembrolizumab — IV infusion

SUMMARY:
An open-label, controlled, multi-site, interventional, 2-arm, Phase II/III trial of BNT113 in combination with pembrolizumab vs pembrolizumab monotherapy as first line treatment in patients with unresectable recurrent or metastatic HPV16+ HNSCC expressing programmed cell death ligand-1 (PD-L1) with combined positive score (CPS) ≥1.

This trial has two parts.

Part A, is an initial non-randomized Safety Run-In Phase to confirm the safety and tolerability at the selected dose range level of BNT113 in combination with pembrolizumab.

Part B, is a randomized part to generate pivotal efficacy and safety data of BNT113 in combination with pembrolizumab versus pembrolizumab monotherapy in the first line setting in patients with unresectable recurrent or metastatic HPV16+ HNSCC expressing PD-L1 with CPS ≥1. Patients included in the Safety Run-In Phase of the trial (Part A) will not be randomized to Part B and will continue on-trial treatment (BNT113 plus pembrolizumab) within Part A.

For Part B, an optional pre-screening phase is available for all patients where patients' tumor samples may be submitted for central HPV16 DNA and central PD-L1 expression testing prior to screening into the main trial.

Patients will be treated with BNT113 in combination with pembrolizumab or with pembrolizumab monotherapy for approximately up to 24 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must sign the written pre-screening informed consent form (ICF) before any pre-screening procedures.
* Patients who present histologically confirmed recurrent or metastatic HPV16+ HNSCC that is considered incurable by local therapies.
* Patients who have a tumor that expresses PD-L1 [CPS ≥1] as determined by the European Conformity (CE)-marked/Food and Drug Administration-approved CDx PD-L1 immunohistochemistry 22C3 pharmDx performed according to the manufacturer's instructions for use.
* Patients must not have had prior systemic anticancer therapy administered in the incurable recurrent or metastatic setting. Systemic therapy which was completed more than 180 days prior to randomization, if given as part of multimodal treatment for locally advanced disease, is allowed.
* Patients who have measurable disease based on RECIST 1.1 as determined by the site and confirmed by BICR. Tumor lesions situated in a previously irradiated area may be considered measurable, if progression has been demonstrated in such lesions disease by RECIST 1.1.
* All patients must provide a tumor tissue sample (formalin fixed paraffin embedded [FFPE] blocks or both slides and curls) from archival tissue. Alternatively, a fresh biopsy sample could be provided if a biopsy sample is performed as part of the patient's standard clinical practice before the first dose of trial treatment. The sample should be preferably derived from a current site of metastatic or recurrent disease. Otherwise, a sample from the primary tumor can be submitted.

Key Exclusion Criteria:

Medical conditions:

* Patients present primary tumor site of nasopharynx (any histology).
* Patients with another primary malignancy that has not been in complete remission for at least 2 years, with the exception of those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, non-invasive basal or non-invasive squamous cell skin cancer, localized prostate cancer, non-invasive superficial bladder cancer or breast ductal carcinoma in situ).

Prior/concomitant therapy:

* Patients who have received or currently receive the following therapy/medication:

  1. Chronic systemic immunosuppressive treatment including corticosteroid treatment (prednisone >10 mg daily orally [PO] or intravenously [IV], or equivalent) in the 7 days prior to the first dose of trial treatment.
  2. Prior treatment with other immune-modulating agents that was (a) within fewer than 4 weeks (28 days) or five half-lives of the agent (whichever is longer) prior to the first dose of BNT113, or (b) associated with immune-mediated AEs that have not resolved prior to the first dose of BNT113 or that pose an additional risk of on-trial complications, per investigator's assessment, or c) associated with toxicity that resulted in discontinuation of the immune-modulating agent and that poses an additional risk of on-trial complications, per investigator's assessment.
  3. Prior treatment with live attenuated vaccines within 4 weeks before the first dose of BNT113.
  4. Prior treatment with an investigational drug (including investigational vaccines) within 4 weeks or five half-lives of the agent (whichever is longer) before the planned first dose of BNT113.
  5. Ongoing treatment with therapeutic PO or IV antibiotics. Note: Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) may be enrolled.
* Prior treatment with anti-cancer immunomodulating agents, such as blockers of programmed death receptor-1 (PD-1), PD-L1, tumor necrosis factor receptor superfamily member 9 (TNRSF9, 4 1BB, CD137), OX 40, therapeutic vaccines, cytokine treatments, or any investigational agent within 4 weeks or five half-lives of the agent (whichever is longer) before the first dose of BNT113.
* Treatment with non-systemic anti-cancer therapy (e.g., radiotherapy or surgery) within 2 weeks prior to randomization. Note: Prior treatment with bone resorptive therapy, such as bisphosphonates (e.g., pamidronate, zoledronic acid) and denosumab, is allowed.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Part A - Occurrence of treatment-emergent adverse event (TEAE) - BNT113 in combination with pembrolizumab | up to 27 months
  TEAE assessed according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) including Grade ≥3, serious, and fatal TEAEs, by relationship.
Part B - Overall survival (OS) | up to 48 months
  OS defined as the time from randomization to death from any cause.
Part B - Progression-free survival (PFS) | up to 48 months
  PFS defined as the time from randomization to the first objective tumor progression (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1] assessed by the blinded independent central review [BICR]), or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Part A and B - Overall response rate (ORR) | up to 48 months
  ORR defined as the proportion of patients in whom a complete response (CR) or partial response (PR) (per RECIST 1.1 assessed by BICR and investigator) is observed as best overall response.
Part A and B - Duration of response (DOR) | up to 48 months
  DOR defined as the time from first objective response (CR or PR per RECIST 1.1) to first occurrence of objective tumor progression (progressive disease [PD] per RECIST 1.1) or death from any cause, whichever occurs first. In Part A, assessment will be done by both BICR and investigator; in Part B, only by BICR.
Part A - Disease control rate (DCR) | up to 48 months
  DCR defined as the proportion of patients in whom a CR or PR or stable disease (SD) (per RECIST 1.1, assessed at least 6 weeks after first dose by BICR and investigator) is observed as best overall response.
Part B - Progression free survival (PFS) | up to 48 months
  PFS defined as the time from randomization to the first objective tumor progression (per RECIST 1.1 by investigator's assessment) or death from any cause, whichever occurs first.
Part B - PFS rate at 6 months | from randomization until 6 months after randomization
  Defined as the proportion of patients without objective tumor progression (per RECIST 1.1 assessed by BICR and investigator) or death from any cause
Part B - PFS rate at 12 months | from randomization until 12 months after randomization
  Defined as the proportion of patients without objective tumor progression (per RECIST 1.1 assessed by BICR and investigator) or death from any cause.
Part B - Occurrence of TEAEs - BNT113 in combination with pembrolizumab compared to pembrolizumab monotherapy | up to 27 months
  TEAEs assessed according to CTCAE v5.0 including Grade ≥3, serious, and fatal TEAEs by relationship.
Part B - Occurrence of dose reduction, delay, and discontinuation of trial treatments due to TEAEs | up to 27 months
  BNT113 in combination with pembrolizumab compared to pembrolizumab monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (189):
- United States (17):
  - California Research Institute, Los Angeles, California
  - UCLA Cancer Care, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - The George Washington Cancer Center, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - The University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - MultiCare Regional Cancer Center, Tacoma, Washington
- Argentina (9):
  - Centro de Oncología e Investigación Buenos Aires COIBA, Berazategui
  - Hospital Britanico de Buenos Aires, Ciudad de Buenos Aires
  - Instituto de Oncologia de Cordoba, Córdoba
  - Centro Oncologico Riojano Integral, La Rioja
  - Centro de Investigacion Pergamino SA - Clinica Pergamino, Pergamino
  - Instituto de Oncologia de Rosario, Rosario
  - Sanatorio Britanico, Rosario
  - CAIPO Centro para la Atencion Integral del Paciente Oncologico, San Miguel de Tucumán
  - Clinica Viedma, Viedma
- Australia (8):
  - Cancer Research SA, Adelaide
  - Bankstown-Lidcombe Hospital, Bankstown
  - Flinders Medical Centre, Bedford Park
  - Coffs Harbour Hospital, Coffs Harbour
  - St Vincent's Hospital, Fitzroy
  - Royal North Shore Hospital, Saint Leonards
  - John Flynn Private Hospital, Tugun
  - Southern Medical Day Care Centre, Wollongong
- Austria (4):
  - LKH - Univ. Klinikum Graz, Graz
  - Landeskrankenhaus/ Univ.-Kliniken Innsbruck, Innsbruck
  - HNO, Kopf-und Halschirurgie Ordensklinikum Linz Barmherzigen Schwestern, Linz
  - Uniklinikum Salzburg, Univ. Klinik fur Innere Medizin III, Salzburg
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent UZ Gent, Ghent
  - CHR de la Citadelle, Liège
- Brazil (13):
  - Fundação PIO XII - Hospital de Amor Barretos, Barretos
  - Fundacao Universidade de Caxias do Sul - Instituto de Pesquisas em Saude IPS-UCS, Caxias do Sul
  - Hospital Erasto Gaertner, Curitiba
  - Oncosite - Centro de Pesquisa Clinica em Oncologia, Ijuí
  - Hospital Marcio Cunha, Ipatinga
  - Irmandade Santa Casa de Misericordia de Porto Alegre Hospital Santa Rita, Porto Alegre
  - Hospital Mae de Deus, Porto Alegre
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto Nacional de Cancer Jose de Alencar Gomes da Silva - INCA, Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto
  - Instituto do Cancer do Estado de São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Cancer, Vila Mariana
- Canada (5):
  - Cross Cancer Institute, Edmonton
  - British Columbia Cancer Agency, Kelowna
  - Jewish General Hospital, Montreal
  - McGill University Health Centre, Montreal
  - Princess Margaret Cancer Centre, Toronto
- Chile (3):
  - Centro de Estudios Clinicos SAGA, Santiago
  - Fundación Arturo López Pérez, Santiago
  - James Lind Centro de Investigación del Cáncer, Temuco
- Czechia (2):
  - Fakultni Nemocnice Olomouc, Olomouc
  - Hospital Na Bulovce (Nemocnice na Bulovce), Prague 8 - Liben
- France (11):
  - CHU de BORDEAUX, Hopital Saint Andre, Bordeaux
  - CHU de Caen Normandie, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Institut de Radiothérapie Hartmann, GCS CCConcorde, Levallois-Perret
  - Hopital de la Timone, Marseille
  - Hopital Prive du Confluent, Nantes
  - Institut Curie, Paris
  - Institut Curie, Groupe Hospitalier Paris Saint-Joseph (GHPSJ), Paris
  - CHU de Tours Hopital Bretonneau, Tours
  - Hospital Gustave Roussy, Villejuif
- Germany (15):
  - Charite Universitätsklinikum Berlin - Campus Benjamin Franklin, Berlin
  - Klinik für HNO-Heilkunde, Kopf- und Hals-Chirurgie, Cologne
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - SRH Wald-Klinikum Gera GmbH, Hamburg
  - Kath. Marien Krankenhaus gGmbH, Hamburg
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitaetsklinik Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - UNIVERSITAETSMEDIZIN der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Klinikum rechts der Isar der TUM, München
  - Univeritätsklinikum Münster, Münster
  - Universitaetsmedizin Rostock - Medizinische Klink III (Hamatologie, Onkologie, Palliativmedizin), Rostock
  - Caritas Klinikum Saarbrucken St. Theresia, Saarbrücken
  - Medizinische Universitaetsklinik Tuebingen, Tübingen
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (4):
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Uzsoki Utcai Korhaz Onkologiai Osztaly, Budapest
  - DEKK Onkologiai Klinika, Debrecen
  - Zala Megyei S. Rafael Korhaz, Zalaegerszeg
- Israel (4):
  - Rambam Health Clinical, Haifa
  - Hadassah Medical Center - Sharett Institute of Oncology, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - ASST Spedali Civili Brescia, Brescia
  - Mater Salutis Hospital AULSS 9 della Regione Veneto, Legnago
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Istituto Europeo di Oncologia, Milan
  - Ospedale del Mare, Napoli
  - A.O.U. Maggiore della Carita, Novara
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
  - Azienda Sanitaria Universitaria Integrata Friuli Centrale - Presidio ospedaliero di Udine, Udine
- Mexico (9):
  - Centro de Estudios y Prevención del Cáncer (CEPREC), Tuxtla Gutiérrez, Region Chiapas
  - Centro Estatal de Cancerologia de Chihuahua, Chihuahua City
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Cryptex Investigacion SA de CV, Mexico City
  - Consultorio del Dr. Joaquín Gabriel Reinoso Toledo, Monterrey
  - Hospital Universitario "Dr Jose Eleuterio Gonzalez" Centro Universitario contra el Cáncer, Monterrey
  - Oaxaca Site Management Organization S. C., Oaxaca City
  - Sociedad de Metabolismo y Corazón S.C., Veracruz
  - Centro de Atencion e Investigacion Clinica en Oncologia (CAICO), Yucatán
- Poland (7):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp.zo.o, Gdynia
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Gliwice
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin
  - MCM Pratia Krakow, Krakow
  - Centrum Medyczne Pratia Poznań, Poznan
  - Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Wroclaw
- Portugal (6):
  - Centro Clinico Academico, Braga
  - Instituto Português de Oncologia de Coimbra Francisco Gentil, E.P.E., Coimbra
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Gaia
  - IPO Lisboa Francisco Gentil, Lisbon
  - Centro Hospitalar Universitario Lisboa Norte, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E, Porto
- South Korea (8):
  - Chungnam National University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - Ajou University Hospital, Suwon
- Spain (12):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Univ. Dr. Josep Trueta, Girona
  - Complejo Hospitalario de Jaen, Jaén
  - Clinica Universidad de Navarra - Madrid (CUN-M), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Regional de Malaga, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Clinica Universidad de Navarra - Pamplona (CUN-P), Pamplona
  - Hospital La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Norrlands University Hospital, Umeå
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Bing Show Chwan Memorial Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital-Kaohsiung Branch, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (12):
  - Medical Park Seyhan Hospital, Adana
  - Hacettepe University Cancer Institute, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Trakya University, Edirne
  - Istanbul Universitesi Onkoloji Enstitusu, Istanbul
  - Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Istanbul
  - Medipol Mega Universite Hastanesi, Istanbul
  - Istanbul Medeniyet University Medical Faculty, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi - Tulay Aktas Onkoloji Hastanesi, Izmir
  - Medical Park - Izmir Hastanesi, Izmir
  - Inonu Universitesi - Turgut Ozal Tip Merkezi, Malatya
  - Baskent University, Yüreğir
- United Kingdom (19):
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast Health and Social Care Trust, Belfast City Hospital, Belfast
  - University Hospitals Birmingham, Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's Hospital - Cambridge University Hospitals, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Teaching Hospitals NHS Trust (St James's University Hospital), Leeds
  - The Clatterbridge Cancer Centre, Liverpool
  - University College London Hospitals, London
  - Guy's Cancer Centre, Guy's Hospital, London
  - The Royal Marsden Hospital NHS Foundation Trust - Fulham Road, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford Cancer Centre, Oxford
  - Royal Preston Hospital Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Mount Vernon Cancer Centre, East and North Hertfordshire NHS Trust, Stevenage
  - The Royal Marsden Hospital - Sutton, Sutton
  - Torbay Hospital - South Devon Healthcare NHS Foundation Trust, Torquay

IPD SHARING:
Plan to Share IPD: No